CLINICAL TRIAL: NCT02009254
Title: The Effect of Mashed Potato Composition on Food Intake, Satiety and Blood Glucose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, G. Harvey Anderson, Professor, University of Toronto
Purpose: Prevention
Other Study IDs: Potato study 2: mashed potato
Record Dates: First submitted 2013-12-08; First posted 2013-12-11 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Obesity; Overweight; Diabetes; Metabolic Syndrome
MeSH Terms: conditions — Obesity; Overweight; Diabetes Mellitus; Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Mashed Potatoes (as produced) (Experimental)
  Interventions: Other: Dietary treatment
- Mashed Potatoes (with no added butter during production) (Experimental)
  Interventions: Other: Dietary treatment
- glucose control (50 g) (Experimental)
  Interventions: Other: Dietary treatment

INTERVENTIONS:
Other: Dietary treatment

SUMMARY:
Potato is one of the world's most popular foods and is widely accepted as a staple food. The objective of this study is to determine the effect of consuming instant mashed potatoes with and without fat on glycemic response, subjective appetite and food intake. It is hypothesized that mashed potato with added fat (as it is usually consumed) will result in lower glycaemic response and subjective appetite, and reduced subsequent food intake.

ELIGIBILITY:
Inclusion Criteria:

* •Healthy men with a body mass index (kg/m2) of 20-24.9

Exclusion Criteria:

* •smocking, medication, breakfast skipping, restrained eating

Ages: 18 Years to 35 Years | Sex: Male
Age Groups: Adult
Dates: Primary Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
blood glucose | 120 min

SECONDARY OUTCOMES:
food intake | 120 min

OTHER OUTCOMES:
subjective appetite | 120 min